CLINICAL TRIAL: NCT05470699
Title: A Prospective Study of the RefleXion [18F]- DCFPyL PET-CT Subsystem Imaging Performance in Patients With Prostate Cancer
Brief Title: RefleXion PET/CT Imaging Performance in Patients With Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22189; NCI-2022-05684 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22189 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic ([18F]-DCFPyL PET-CT, X1 RMRS PET-CT) (Experimental): Patients receive [18F]-DCFPyL IV and undergo [18F]-DCFPyL PET-CT over 30 minutes per SOC. Patients with PET avid lesions then undergo a X1 RMRS PET-CT imaging-only session within 120 minutes of injection over 20-35 minutes.
  Interventions: Procedure: Computed Tomography; Other: Fluorine F 18 Piflufolastat; Device: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Other: Fluorine F 18 Piflufolastat — Given IV
  Other Names: 18F-DCFPyL; Fluorine F 18 DCFPyL; Piflufolastat F 18; Piflufolastat F-18; Piflufolastat F18; Pylarify
Device: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This clinical trial examines RefleXion Medical Radiotherapy System (RMRS) imaging to the standard of care (SOC) [18F]-DCFPyL positron emission tomography-computed tomography (PET-CT) imaging in patients with prostate cancer. PET is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of a tracer, [18F]-DCFPyL, that binds to prostate specific membrane antigen (PSMA) on tumor cells. These PSMA tumor cells can then be identified on PET imaging. CT utilizes x-rays that traverse body from the outside. CT images provide an exact outline of organs and potential inflammatory tissue where it occurs in patient's body. The RMRS is a imaging-therapy combination system that can plan for and deliver radiation therapy as well perform [18F]-DCFPyL PET-CT imaging. Comparing the imaging from the standard of care [18F]-DCFPyL-PET-CT with the [18F]-DCFPyL imaging from RMRS may help improve the quality of the imaging captured and determine if imaging can be done on the RMRS at the same time as planning for radiation therapy, which would reduce the number of scans needed to plan for radiation for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess imaging performance of the fluorine F 18 piflufolastat ([18F]-DCFPyL) PET-CT subsystem on the X1 RMRS to detect lesions (primary and metastatic) in patients with prostate cancer.

SECONDARY OBJECTIVE:

I. To determine the feasibility of generating a biology-guided radiotherapy (BgRT) plan using X1 RMRS-acquired [18F]-DCFPyL PET data derived from the imaging-only session at the studied dose level.

OUTLINE:

Patients receive [18F]-DCFPyL intravenously (IV) and undergo [18F]-DCFPyL PET-CT over 30 minutes per standard of care (SOC). Patients with PET avid lesions then undergo a X1 RMRS PET-CT imaging-only session within 120 minutes of injection over 20-35 minutes.

After completion of study, patients are followed up within 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Age >= 21 years
* Patients undergoing SOC [18F]-DCFPyL PET-CT
* Patients should be scheduled for [18F]-DCFPyL PET-CT prior to study entry

Exclusion Criteria:

* Known psychiatric or substance abuse disorder that would interfere with conduct of the study
* Patient weight exceeding the weight limit (450 pounds) outlined per X1 RMRS specifications sheet

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2026-04-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Y Wong, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 34 patients provided informed consent.
Period: Overall Study
Arm/Group | Diagnostic ([18F]-DCFPyL PET-CT, X1 RMRS PET-CT)
Started | 34
Completed | 20
Not Completed | 14
Not completed — Did not receive intervention | 13
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic ([18F]-DCFPyL PET-CT, X1 RMRS PET-CT)
Number analyzed (Participants) | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72 [63 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 11
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Tumor Visualized on X1 RefleXion Medical Radiotherapy System (RMRS) Positron Emission Tomography-computed Tomography (PET-CT)
Description: To determine imaging performance of the X1 PET scan, the number of tumors clearly visualized on PET scan were reported.
Time Frame: Up to 72 hours after completion of scan
Population: Biology-guided radiotherapy plans were successfully generated for 18 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic ([18F]-DCFPyL PET-CT, X1 RMRS PET-CT)
Number analyzed (Participants) | 18
Participants | 1

2. Secondary Outcome: Percent of Cases Where X1 RMRS [18F]-DCFPyL PET Data Can be Used to Generate an Acceptable Biology-guided Radiotherapy (BgRT) Plan
Description: The true positive lesions identified on the X1 PET images will be identified and used for BgRT planning. Simulated planning using the RefleXion treatment planning software will be performed, and the radiation dose to organs at risk calculated. Principal investigator will determine whether this plan is acceptable or not. The percent of cases in which RefleXion [18F]-DCFPyL PET data led to an acceptable plan will be recorded (descriptive statistics). Descriptive statistics will be utilized to quantify results. Mean, standard deviation, IQR, and range will be reported for each continuous variable. Frequency and percentage will be reported for categorical variables. Statistical significance will be assessed at the 0.05 level, one-sided.
Time Frame: Up to 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic ([18F]-DCFPyL PET-CT, X1 RMRS PET-CT)
Number analyzed (Participants) | 20
Participants | 18

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the beginning of the imaging-only session on the X1 RMRS system and continued until 72 hours after the end of the scan.
Arm/Group | Diagnostic ([18F]-DCFPyL PET-CT, X1 RMRS PET-CT)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 4/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic ([18F]-DCFPyL PET-CT, X1 RMRS PET-CT) (N=20)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT05470699/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT05470699/ICF_001.pdf